CLINICAL TRIAL: NCT01426334
Title: Exploiting Synergy in Chronic Myelogenous Leukemia: A Phase Ib Evaluation of Dasatinib Plus Cyclosporine in Patients With Ph+ Leukemia (ESCAPE1b)
Brief Title: Dasatinib and Cyclosporine in Treating Patients With Chronic Myelogenous Leukemia Refractory or Intolerant to Imatinib Mesylate
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-03454; NCI-2011-03454 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000709681; 10-1401; 10-1401 (Other: University of Colorado Cancer Center - Anschutz Cancer Pavilion); 8890 (Other: CTEP); P30CA046934 (NIH); NCT01456988 (obsolete NCT alias)
Record Dates: First submitted 2011-08-30; First posted 2011-08-31 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2013-06

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia; Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Chronic Phase Chronic Myelogenous Leukemia; Relapsing Chronic Myelogenous Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Chronic-Phase | interventions — Dasatinib; Cyclosporine

ARMS (1):
- Treatment (dasatinib and cyclosporine) (Experimental): Patients receive dasatinib PO QD on days 1-28 and cyclosporine PO BID on days 8-28. Treatment repeats every 28 days for 4 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: dasatinib; Other: diagnostic laboratory biomarker analysis; Other: pharmacological study; Drug: cyclosporine

INTERVENTIONS:
Drug: dasatinib — Given PO
  Other Names: BMS-354825; Sprycel
Other: diagnostic laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Drug: cyclosporine — Given PO
  Other Names: ciclosporin; cyclosporin; cyclosporin A; CYSP; Sandimmune

SUMMARY:
This phase I trial studies the side effects and the best way to give dasatinib and cyclosporine in treating patients with chronic myelogenous leukemia (CML) refractory or intolerant to imatinib mesylate. Dasatinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Cyclosporine may help dasatinib work better by making cancer cells more sensitive to the drug. Giving dasatinib together with cyclosporine may be an effective treatment for CML.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To define the safety and tolerability of cyclosporine A in combination with dasatinib in adults with Bcr-Abl+ chronic myelogenous leukemia in chronic phase, or when used in specified patients with accelerated phase CML.

SECONDARY OBJECTIVES:

I. To assess pharmacokinetic parameters of dasatinib when combined with cyclosporine.

II. To assess whether the combination of dasatinib and cyclosporine alters T cell number and function.

III. To assess the feasibility of determining phosphorylation of Src in peripheral blood mononuclear cells by flow cytometry as a surrogate measure of dasatinib activity.

OUTLINE:

Patients receive dasatinib orally (PO) once daily (QD) on days 1-28 and cyclosporine PO twice daily (BID) on days 8-28. Treatment repeats every 28 days for 4 months in the absence of disease progression or unacceptable toxicity.

Patients undergo peripheral blood sample collection at baseline and periodically during treatment for pharmacokinetic and pharmacodynamic studies and T-cell number and function by flow cytometry.

After completion of study treatment, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed chronic myelogenous leukemia (CML), Philadelphia chromosome positive (Ph+)
* Patients must have a diagnosis of:

  * de novo chronic phase Ph+ CML, and not have received therapy with a tyrosine kinase inhibitor (TKI) for more than 2 weeks prior to enrollment
  * OR chronic phase Ph+ CML refractory to or with intolerance of treatment with imatinib or nilotinib therapy; patients being treated with dasatinib who have refractory disease may be considered for inclusion, at the discretion of the PIs, if other therapeutic options are not deemed likely to be efficacious (e.g. previous intolerance or refractoriness to nilotinib); evaluation for and consideration of hematopoietic stem cell transplantation as appropriate to the patient's condition by the patient's primary treating hematologist/oncologist should occur prior to enrollment in this trial
  * OR chronic phase Ph+ CML, without complete molecular remission after 3 months of treatment with imatinib, nilotinib or dasatinib
  * OR accelerated phase Ph+ CML, for which allogeneic hematopoietic stem cell transplantation is being planned, and for which no cytotoxic chemotherapy is planned prior to conditioning, and can be reasonably expected to participate for a minimum of one month prior to transplantation
  * OR accelerated phase Ph+ CML, for which allogeneic hematopoietic stem cell transplantation is not a therapeutic option (due to age or lack of acceptable donor, for example), and can be reasonably expected to participate for a minimum of one month
* Chronic phase CML shall be defined by the presence of fewer than 15% blasts, fewer than 20% basophils, and fewer than 30% blasts plus promyelocytes in the peripheral blood and bone marrow, no extramedullary involvement except liver and spleen, and no evidence of clonal evolution (O'Brien et al., 2003)
* Treatment failure/refractory disease shall be defined as less than complete hematologic response at 3 months, no cytogenetic response at 6 months, less than partial cytogenetic response at 12 months, less than complete cytogenetic response at 18 months, OR loss of CHR, loss of CCyR, clonal chromosomal abnormalities, detection of imatinib insensitive mutations, or 1 log increase in BCR-ABL transcript level from best molecular response documented on 2 samples at least one month apart (Baccarani et al., 2009)
* Intolerance of TKI therapy shall be defined by non-hematologic toxic effects of any grade leading to intermittent or chronic non-compliance with, repeated dose reduction or delays in continuous dosing, or discontinuation of Imatinib
* Accelerated phase CML shall be defined as the presence of >= 15-29% blasts, >= 20% basophils, or >= 30% blasts plus promyelocytes in the peripheral blood or bone marrow, thrombocytopenia unrelated to therapy, or evidence of cytogenetic clonal evolution (Kantarjian et al., 1993)
* Prior Therapy

  * Patients must have discontinued imatinib, nilotinib or dasatinib at least 7 days prior to starting study therapy; this washout period may be omitted at the discretion of the PIs, if it is determined that the washout may adversely affect patient care
  * Patients must discontinue hydroxyurea or interferon at least 7 days prior to starting study therapy
* Life expectancy of greater than 1 month
* ECOG performance status =< 2 (Karnofsky >= 60%)
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,000/mcL
* Absolute CD4+ count >= 350/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within normal institutional limits
* AST(SGOT)/ALT(SGPT) =< 2.5 X institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* The effects of dasatinib on the developing human fetus are unknown; for this reason and because PTK inhibitors are known to be teratogenic, women of childbearing potential must have a negative pregnancy test within 7 days of study entry; women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and for a minimum of 30 days following discontinuation of study therapy; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; lactating women must agree not to nurse a child while on this trial or within 30 days of discontinuation of study therapy
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or failure to recover from adverse events (except alopecia) to Grade =< 1 or to baseline (if there is persistent, chronic, stable Grade 2), due to agents administered more than 4 weeks earlier
* Patients may not be receiving any other investigational agents
* Known brain metastases exclude patients from this clinical trial because such patients have a poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events; in addition, patients who have active brain metastases may benefit from other concurrent therapy such as radiation or radiosurgery, and should be considered for the most appropriate clinical therapy that may provide symptom relief
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to dasatinib or cyclosporine
* Patients who require concurrent treatment with any medications or substances that are potent inhibitors or inducers of CYP3A4 are ineligible; efforts should be made to switch patients with a seizure disorder who are taking enzyme-inducing anticonvulsant agents to other medications
* Patients who require concurrent treatment with proarrhythmic potential
* QTc prolongation (defined as a QTc interval >= 480 msec) or other significant ECG abnormalities
* Use of antithrombotic and/or anti-platelet agents (e.g., warfarin, heparin, low molecular weight heparin, aspirin, and/or ibuprofen); exception: patients with CML who have significantly elevated platelet counts taking anagrelide are eligible; patients who require < 2 mg of warfarin per day for central venous catheter prophylaxis are allowed on this study
* Patients with any condition (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease) that impairs their ability to swallow and retain dasatinib tablets are excluded; tablets may not be crushed prior to administration
* Patients may not have any clinically significant cardiovascular disease, defined as NYHA class III or higher and as follows:

  * Myocardial infarction or ventricular tachyarrhythmia within 6 months
  * Prolonged QTc >= 480 msec (Fridericia correction)
  * Ejection fraction less than institutional normal
  * Major conduction abnormality (unless a cardiac pacemaker is present)
* Patients with any cardiopulmonary symptoms of unknown cause (e.g. shortness of breath, chest pain, etc.) should be evaluated by a baseline echocardiogram with or without stress test as needed in addition to electrocardiogram (EKG) to rule out QTc prolongation; the patient may be referred to a cardiologist at the discretion of the principal investigator; patients with underlying cardiopulmonary dysfunction should be excluded from the study
* Uncontrolled intercurrent illness including, but not limited to, the following: ongoing or active infection; history of significant bleeding disorder, including congenital (von Willebrand's disease) or acquired (anti-factor VIII antibodies) disorders; large pleural effusions; or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because animal studies with dasatinib have shown embryolethality and fetal skeletal alterations at non-toxic maternal doses; because there is an unknown but potential risk for adverse events in nursing human infants secondary to treatment of the mother with dasatinib, breastfeeding should be discontinued if the mother is treated with dasatinib
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with dasatinib; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated
* Known congenital or acquired immunodeficiency
* CD4+ count less than 350/µl
* Mutation in Bcr-Abl known to confer resistance to dasatinib; (N.B. patients for whom Bcr-Abl mutations have not been assessed, will have this assessment in screening; they will be allowed to enroll and initiate therapy; if screening analysis reveals Bcr-Abl mutation known to confer resistance to dasatinib, the patient will be discontinued from study participation)
* Prior hematopoietic stem cell transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-09; Primary Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of combining dasatinib and cyclosporine, as assessed by the incidence of adverse events and serious adverse events in this patient population | Up to 4 weeks post-treatment
  Serious adverse events, toxicity, and patient withdrawals/discontinuations will be determined by the severity, duration, causality, seriousness, and type of event as defined in the protocol.

SECONDARY OUTCOMES:
Pharmacokinetic profiles of patients taking dasatinib alone versus dasatinib with cyclosporine | At baseline and on days 7, 21, 49, 77, and 105
  Exposure to dasatinib will be determined and compared using peak levels (Cmax) and areas under the curve (AUC). Paired t-tests will be used to determine statistical significance.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Porter, Principal Investigator — University of Colorado Cancer Center - Anschutz Cancer Pavilion
Locations (2):
- United States (2):
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - University of Colorado, Denver, Colorado